CLINICAL TRIAL: NCT04452396
Title: Continuous Glucose Monitoring: An Evaluation of Impact on Improving the Efficiency of Diagnostic Processes and Enhancing Patient Safety in the Management of Reactive and Spontaneous Hypoglycaemia
Brief Title: CGM (Continuous Glucose Monitoring) Use in Diagnosis of Spontaneous and Reactive Hypoglycaemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the Covid crisis: clinical changes in staff, bed pressures and time restraints.
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 265405
Record Dates: First submitted 2019-11-18; First posted 2020-06-30 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Hypoglycemia, Reactive; Hypoglycaemia Night; Hypoglycemia Non-Diabetic; Hypoglycemia Unawareness; Insulinoma; Insulinoma; Malignant, Pancreas; Insulin Hypoglycemia; Insulin Resistance; Spontaneous Hypoglycemia; Neuro Endocrine Tumours
Keywords: hypoglycaemia; insulinoma
MeSH Terms: conditions — Hypoglycemia; Insulinoma; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: 2 phases to study. Patients can enter at start of either phase and start phase 2 at the end of phase 1.
  Phase 1 - CGM monitoring of people with suspected spontaneous/reactive hypoglycaemia phase 2 - CGM monitoring of patients with medically managed spontaneous/reactive hypoglycaemia
Masking Description: Phase 1 - (diagnostic) The CGM device will be blinded to the patient and physician until investigations into hypoglycaemia are complete phase 2 - (treatment optimisation) The CGM device will be blinded to the patient and physician for the first 10 days of treatment, medication will be optimised and the patient will continue with CGM in an unblinded way for up to 20 further days to aid further treatment optimisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): patients undergoing CGM monitoring
  Interventions: Device: use of continuous glucose monitoring

INTERVENTIONS:
Device: use of continuous glucose monitoring — Patients will wear a CGM device whilst undergoing diagnostic testing for reactive/spontaneous hypoglycaemia and then optimisation of anti-hypoglycaemic medication.

SUMMARY:
Use of CGM to determine diagnosis in possible spontaneous or reactive hypoglycaemia.

Use of CGM to aid treatment optimisation in spontaneous or reactive hypoglycaemia

DETAILED DESCRIPTION:
The human body's blood sugar levels are tightly controlled by the hormone insulin, produced by the pancreas. If the pancreas produces too much insulin, then the blood sugar will fall to low levels (hypoglycaemia). Insulin overproduction can happen as a result of the body misreading a change in blood sugar levels after eating (such as after obesity surgery) or through tumours of the pancreas which overproduce insulin (insulinomas).

Hypoglycaemia can cause subtle symptoms such as tiredness, poor concentration, or dizziness and if untreated more severe symptoms including fits, coma and death. Low blood sugars can go unnoticed at night and if levels fall frequently, people can lose their ability to notice subtle symptoms.

People suspected of having hypoglycaemia require a series of investigations to try and reproduce a low blood sugar under controlled conditions. This often requires an admission to hospital for a few days and multiple finger pricks to test the blood sugar - which patients often find painful. If low blood sugars caused by too much insulin are confirmed then medical treatment is started in the first instance, with surgery possibly following later. The only way to check whether these medications are working is by home fingerprick glucose measurements. If people have low sugars at night or have lost their ability to notice symptoms of low blood sugar, it is very difficult to be sure that the medical treatment is working.

The investigators plan to use continuous glucose monitoring probes to measure patient's blood sugar prior to and during admission for formal investigation for hypoglycaemia (alongside conventional fingerprick and blood testing). This might allow us to exclude hypoglycaemia as a cause of their symptoms, avoiding lengthy admissions.

The investigators will also use this technology (alongside fingerprick testing) to test how well medical treatment is working in patients with proven hypoglycaemia.

ELIGIBILITY:
Inclusion Criteria:

* phase 1 - under investigation for possible/probable hypoglycaemia
* phase 2 - on medical therapy for established hypoglycaemia
* Must be Able and willing to give informed consent. No vulnerable adults will be included.
* Must be Aged >18 years

Can be;

* Any ethnicity
* Any socio economic group
* Either conventional gender, or non-binary.

Exclusion Criteria:

* Must not be unwilling or unable to give consent
* Must not be unable to speak sufficient English to give consent and understand study requirements
* Must not be Aged<18 or >90 years
* Must not be lack capacity to consent
* Must not have an underlying hepatic condition
* Must not have a current excessive alcohol consumption (men regularly consuming >50 units/week, women >35 units/week)
* Must not have Diabetes Mellitus
* Must not be currently using Diabetic medication or insulin
* Must not be currently pregnant
* Must not be on haemo or peritoneal dialysis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
study arm 1 - diagnosing hypoglycaemic episodes using Continuous Glucose Monitoring of interstitial fluid as a proxy marker of blood glucose | up to 5 days prior to admission for hypoglycaemia investigations
  outpatient - CGM findings reflect patient's fingerprick glucose readings
  * Episodes of true hypoglycaemia (glucose measurement <4, <3.0, <2.2mmol/L as decided by finger prick glucose testing) are captured by the CGM device
study arm 1 - diagnosing hypoglycaemic episodes (glucose measurement <4mmol/L) using Continuous Glucose Monitoring of interstitial fluid as a proxy marker of blood glucose | up to 5 days in hospital during investigations for hypoglycaemia
  inpatient - CGM findings reflect patient's fingerprick glucose readings
  * Episodes of true hypoglycaemia (glucose measurement <4, <3.0, <2.2mmol/L, as decided by finger prick glucose testing) are captured by the CGM device Inpatient - 72 hour fast - CGM device calls hypoglycaemia (glucose measurement <4, <3.0, <2.2mmol/L) when fingerprick/lab glucoses also do
study arm 2 - using Continuous Glucose Monitoring of interstitial fluid as a proxy marker of blood glucose to optimise hypoglycaemia treatment in patients with an established diagnosis of spontaneous or reactive hypoglycaemia | up to 30 days
  blinded phase - CGM findings reflect patient's fingerprick glucose readings- any episodes of true hypoglycaemia (as decided by fingerprick glucose testing) are captured by CGM device unblinded phase - CGM recordings help with titration of anti hypoglycaemic medications and this reduces overall incidence of hypoglycaemic episodes or duration of time spent in hypoglycaemic range (<4, <3.0, <2.2 mmol/L)

SECONDARY OUTCOMES:
assessing concordance between CGMS and lab/finger prick glucose testing | up to 10 days (study arm 1) or up to 30 days (study arm 2)
  To determine whether CGM systems accurately record hypoglycaemia and can be used in this context

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, dept of endocrinology, London, United Kingdom

DOCUMENTS (2):
  • Study Protocol (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT04452396/Prot_000.pdf
  • Informed Consent Form (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT04452396/ICF_001.pdf